CLINICAL TRIAL: NCT00595569
Title: Flexible, Intensive Insulin Management in Patients With Type 1 Diabetes and Changes in Metabolic Control, Quality of Life, Locus of Control and Diabetes Knowledge
Brief Title: Flexible, Intensive Insulin Therapy in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Diabetes Association Basel (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Dr. Jardena Puer, University of Lausanne Hospitals
Other Study IDs: 120/04; 120/04
Record Dates: First submitted 2007-12-28; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: flexible insulin therapy; diabetes education; diabetes; insulin; Weekly ambulatory sessions
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 diabetes
  Interventions: Behavioral: Flexible insulin therapy (FIT)

INTERVENTIONS:
Behavioral: Flexible insulin therapy (FIT) — Flexible insulin therapy (FIT) courses consisting in 7 weekly ambulatory sessions lasting 90 minutes each

SUMMARY:
To prospectively evaluate the long term metabolic and psychological effects of flexible intensive insulin therapy (FIT) courses in an unselected population of type 1 diabetic patients at the University of Basel Hospital. We hypothesize that both metabolic control and psychological parameters will improve.

ELIGIBILITY:
Inclusion Criteria:

* All patients participating in 5 consecutive FIT courses that began between April 2002 to April 2004

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with type 1 diabetes followed at the Division of Endocrinology and Diabetology, University of Basel are strongly encouraged to attend the course 6 to 12 months after having been diagnosed. The population that participates in those FIT courses includes patients from the University of Basel Hospital, but also patients that are referred from out of hospital physicians/diabetologists.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2002-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Metabolic control (HbA1c, severe hypoglycemic events), psychological effects, diabetes knowledge | Over 18 months

SECONDARY OUTCOMES:
Changes in insulin doses, changes in weight | Over 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jardena J Puder, MD, Principal Investigator — University of Lausanne, University of Basel
Locations (1):
- University of Basel Hospital, Basel, Switzerland